CLINICAL TRIAL: NCT05802719
Title: Study of the Functional Status Neutrophils in Rheumatoid Arthritis Patients to Identify New Biomarkers of Response to Anti-TNFalpha Therapy
Acronym: NeutroARTherap
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL22_0150
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Immunology and Immunotherapy; neutrophils; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Exploratory pathophysiological cohort study, with a prospective 6-months follow-up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rheumatoid arthritis patient (Experimental): patient with an active Rheumatoid arthritis and an indication to start an anti-TNFa treatment
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — The procedure consists of collecting 4 additional tubes of blood (20mL) at each visit for research purposes, in order to perform the immunological assays.
  Blood samples at the inclusion, 3 month and 6 month after initiation of anti-TNF therapy

SUMMARY:
The goal of this interventional pathophysiological exploratory, cohort, prospective, with a 6-month follow-up study is to characterize phenotypic and functional alterations of PolyMorphonuclear Neutrophils as well as monocytes/macrophages and dendritic cells in blood samples from rheumatoid arthritis patients. Investigators will perform prospective characterization of these myeloid cells before and after treatment to assess how the functional status of PMNs/myeloid cells affects the response to anti-TNFα (tumor necrosis factor alpha) in rheumatoid arthritis.

This will identify key immune components potentially involved in the activation and/or recruitment of PolyMorphonuclear Neutrophils (PMN) (and other myeloid cells) that may play a role in the pathogenesis of Rheumatoid Arthritis and may help predict the response to anti-TNFα agents, thus guiding the decision-making of therapeutic strategies.

DETAILED DESCRIPTION:
Rheumatoid Arthritis (RA) is a chronic disease with substantial impact on the lives of millions of people across Europe. It is a disease of considerable socioeconomic burden, with direct and indirect costs across Europe reaching hundreds of billions of Euros per year. Demographic studies indicate that the next decade will see this burden dramatically rise. Ultimately, RA results in substantial pain, disability, adverse social consequences and significantly increased risk of mortality for the individual, while at the same time having a massive impact on health economies across Europe. In recent years, RA treatment has been partially effective due to the introduction of effective, although extremely costly, bDMARDs (biological Disease Modifying Anti-Rheumatic Drug) as monoclonal antibody (mAb)-based therapies.

From the clinical, immunological and molecular perspectives, RA is a heterogeneous disease and treatments effective for one patient frequently do not work for another. Due to individual differences, the response rate to first line treatment currently lies at an inadequate 60-70%. In addition, even if patients with RA frequently achieve an inactive disease status, sustained remission without need of medication is still elusive for most. Considering that mAb-based therapies are still very expensive, it is important to thoroughly identify the mechanisms that block their efficacy as well as the predictive factors of therapeutic response. Thus, a better use of mAb-based therapies could result in a therapeutic benefit but also in a considerable economic reduction for National Health Care Systems.

Most studies of immune cells in RA have limitations, such as the analysis of only a small number of cell subsets (in which PMN are most often not included) and limited integrative longitudinal data on patient phenotypes. Studies on PMN and other myeloid cells activation may lead to the identification of mechanisms of disease induction and maintenance.

It has been described that PMN play diverse roles in various infectious and inflammatory diseases, making them a potentially attractive target for therapeutic intervention. Excessive or inappropriate activation of PMN likely contributes to tissue damage in inflammatory disorders. In such cases, therapeutic neutrophil-targeted strategies should aim to inhibit the neutrophil compartment, either by reducing the number of PMN or by inhibiting their functional response. The latter can be achieved by reducing neutrophil activation or dampening the effects of neutrophil-derived mediators. A number of ongoing studies are therefore aiming to manipulate neutrophils for the treatment of several diseases, with therapeutic approaches including targeting neutrophil development and production, interfering with neutrophil accumulation at the site of infection or inflammation and reversing the detrimental changes of neutrophil phenotype that occur during certain pathological conditions. In the past, drug development efforts have always shied away from targeting PMN, mainly for fear of severe infectious complications. Several studies suggest the existence of a therapeutic window of attenuating neutrophil-mediated inflammatory processes without interfering with neutrophil-mediated host defense. It is possible to envision the development of agents that can block defined neutrophil functions while only modestly impairing host-defense. Therefore, the knowledge gathered about the role of PMN in health and disease will lead to the development of therapeutic strategies that target specific features of PMN biology.

The study of PMN in inflammatory diseases has recently brought the concept of neutrophil heterogeneity and plasticity, which is suggested to occur in a context-dependent manner. Upon specific inflammatory conditions PMN are able to change their phenotypes and molecular properties. However, the phenotypic and functional diversity of PMN is ill-understood in RA pathogenesis and mostly overlooked in response to current treatments, including those involving mAbs. Studying the neutrophil heterogeneity has significant therapeutic relevance. In particular, the identification and characterization of PMN subsets will allow targeting a specific PMN subpopulations with deleterious functions, mitigating their harmful aspects without compromising host defense. It will also be possible to reinforce PMN subsets displaying beneficial functions.

It is worth to mention that until recently, PMN were thought to belong to a relative homogeneous population of cells. However, an increasing number of studies now show heterogeneity in morphology, phenotype, function, or a combination of these factors, particularly in various diseases including RA. However, it is still unclear whether those populations represent different states of a continuous polarization spectrum or reflect other features of the PMN compartment with intrinsic functional differences. In human, one of the subtypes of PMN identified is the low-density neutrophil (LDN). It was first recognized when PMN co-segregated with mononuclear cells after density-gradient isolation in systemic lupus erythematosus (SLE) and RA patients. However, the pathophysiological role of these cells low-density cells is unclear, especially in the context of RA. Low-density granulocytes (LDGs) are heterogeneous and might represent immature and partially degranulated neutrophils that behave differently depending on the disease or, possibly, even a pathological subset of neutrophils that have not differentiated properly. Whether LDGs are a cause or a consequence of disease is unknown.

Several studies have used whole-blood transcriptomics to search for potential biomarkers to predict response to biologic agents in RA, but there is no clear correlation among data from different studies, and no candidate biomarker has progressed to a clinical diagnostic. In addition, transcriptomic studies involving PMN are scarce. Wright and collaborators investigated the profile transcriptome of purified peripheral blood neutrophils from RA patients in response to anti-TNFa treatment. However, this study was performed using preparations of total PMN with no distinction of PMN subsets. Thus, the biological/pathobiological roles of the heterogenous neutrophil subpopulations (including LDG) remains to be elucidated. Similarly, whether and how PMN might modulate the properties of other myeloid cells in RA patients are still underexplored.

Taking into consideration the clinical unmet need and the therapeutic perspectives, our objective is to study the phenotypic and functional alterations in PMN and myeloid cells in RA patients. While available transcriptomic data are informative, data on protein secretion as well as on functional activation are needed to further dissect neutrophil function/dysfunction in RA patients. In this context, investigators will adopt a unique approach to characterize properties of PMN (and subsets) and myeloid subpopulations.

Answering this question may have important implications for the designing of new targeted therapies that influence dysregulated neutrophil function and/or neutralize factors that promote neutrophilic inflammation or their interaction with pathogenic immune cell subsets (as monocytes). It may also improve the management of RA patients by current therapies by helping to give the right drug to the right patient.

Despite progress in the field needs remain unmet, not least in the current absence of the capacity to predict, prevent and cure the disease, but even in the prediction of which patients respond to a particular therapy. It is clear that our Neutro-ARTherapy objectives comply with the perspective of better understanding pathogenetic mechanisms involved in RA, in turn increasing our knowledge in the field and ultimately leading to the discovery of biological therapeutic agents with a more precise decision-making and medicine-based therapeutic prescription.

ELIGIBILITY:
Inclusion Criteria:

* Established RA patients fulfilling 2010 ACR/EULAR (American College of Rheumatology / European League Against Rheumatism) definition Active disease (DAS28 score (Disease Activity Score) > 3.2)
* Indication to start an anti-TNFalpha treatment : adalimumab or etanercept
* 18 years old or older

Exclusion Criteria:

* Current treatment or within 12 months prior to inclusion with Rituximab
* Current treatment or within 1 month prior to inclusion with corticosteroids >10 mg/day (oral or intravenous)
* Contra-indication to TNF inhibitors (active infections, cancer in the last 5 years, active tuberculosis, hepatitis B or C or HIV positive except for hepatitis B vaccination)
* Severe intercurrent inflammatory disease
* Patient unable to give consent : under guardianship, curators or safeguard of justice;
* Pregnant, parturient or nursing woman.
* Participation in an interventional clinical trial
* Patient refusing to give oral informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
The difference in numbers/functional status of PMN (frequency) | Between baseline and 3 months after the initiation of anti TNFa
  The difference in numbers/functional status of PMN between baseline and 3 months post-treatment and related to the DAS28 EULAR response.
  The biomarkers of interest is frequency of PNM after stimulation by inflammatory factors.
The difference in numbers/functional status of PMN (phenotypic properties/activation) | Between baseline and 3 months after the initiation of anti TNFa
  The difference in numbers/functional status of PMN between baseline and 3 months post-treatment and related to the DAS28 EULAR response.
  The biomarkers of interest is phenotypic properties/activation of PMN after stimulation by inflammatory factors.
The difference in numbers/functional status of PMN (in vitro PMN secretory profile) | Between baseline and 3 months after the initiation of anti TNFa
  The difference in numbers/functional status of PMN between baseline and 3 months post-treatment and related to the DAS28 EULAR response.
  The biomarkers of interest is in vitro PMN secretory profile after stimulation by inflammatory factors.

SECONDARY OUTCOMES:
To assess how the frequency and activation of myeloid cell subpopulations in the peripheral blood affects the 3-months clinical response to anti-TNFa therapy | 3 months after the initiation of anti TNFa
To assess how the frequency and activation of myeloid cell subpopulations in the peripheral blood affects the 6-months clinical response to anti-TNFa therapy | 6 months after the initiation of anti TNFa
To assess if the PMN profile varies between baseline and 3 months after initiation of anti-TNFa therapy | between baseline and 3 months after initiation of anti-TNFa therapy
To assess if the PMN profile varies between baseline and 6 months after initiation of anti-TNFa therapy | between baseline and 6 months after initiation of anti-TNFa therapy
To assess if the myeloid cell subpopulations varies between baseline and 3 months after initiation of anti-TNFa therapy | between baseline and 3 months after initiation of anti-TNFa therapy
To assess if the myeloid cell subpopulations varies between baseline and 6 months after initiation of anti-TNFa therapy | between baseline and 6 months after initiation of anti-TNFa therapy
Compare evolution of PMN activity between EULAR responders and non-responders after 6 months of anti-TNFa therapy according to their functional status | After 6 months of anti-TNFa therapy

CONTACTS AND LOCATIONS:
Overall Officials: Christian JORGENSEN, MD PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Centre Hospitalier Universitaire de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No